CLINICAL TRIAL: NCT04335500
Title: Self-reported Fear of Intraoral Injections and Its Relationship to Dental Fear and Subsequent Avoidance of Dental Treatment Among 8 to 10 Years Children: Across Sectional Study
Brief Title: Prevalance of Intraoral Injection Fear
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Mohamed Mosaad Hussien, Principle investigator, Resident at pediatric dentistry department Nora Mohamed Mosaad, Cairo University
Other Study IDs: Inraoral injection fear
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Injection Fear, Fear, Avoidance, Dental
MeSH Terms: conditions — Iatrophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the study

1. Estimate the prevalence of intraoral injection fear and its relationship to dental fear among 8-10 years children.
2. Explore the possible consequences of such problems in terms of avoidance of dental and medical care.

DETAILED DESCRIPTION:
Statement of the problem Despite all the technological advancements in the dental profession, fear toward dentistry remains a major concern and potentially distressing problem in daily practice (Oliveira et al. 2014).

Dental fear is a normal emotional reaction to one or more specific threatening stimuli within the dental situation and Intra oral injection is considered one of the most fear-provoking stimuli in the dental setting. Excessive or unreasonable fear or anxiety can influence daily living and result in prolonged avoidance of dental treatment leading to a public health dilemma (Shim et al. 2015).

People with high dental fear, children and adults, may prove difficult to treat, require more time, and present with behavioral problems which can result in a stressful and unpleasant experience for both the patient and treating dental practitioner (Armfield & Heaton 2013).

Rationale Intra-oral injections have been shown to be among the most fear-provoking stimuli in the dental setting.(Berge et al. 2016) Dental patients with fear and anxiety may also become dependent on pharmacological approaches for the management of their care, particularly if they do not receive treatment for their anxiety (MCGoldrick et al. 2001).

Assessment of high intra-oral injection fear is of paramount impact in offering the affected patients appropriate treatment , such as cognitive behavioral therapy and applied tension. (Berge et al. 2016) Cognitive Behavioral Therapy (CBT) is a goal-orientated talking therapy which aims to help people manage their problems by changing how they think and behave in relation to their problems. CBT incorporates a variety of different cognitive and behavioral strategies which aim to help the patient modify the unhelpful behaviors or thoughts maintaining their anxiety. (Marshman et al. 2018) Applied tension is a treatment method that is used with patients with blood-injection-injury phobia to alter their physiological response to the feared stimulus. The method includes repeated muscle tensing when in the presence of feared stimuli to counteract the drop in blood pressure and prevent vasovagal syncope.(Mednick et al. 2012) During Dental Procedures Some children may experience vasovagal syncope, proper history taking from those patients will help the dentist get prepared for such a probability.(Vika et al. 2008) Some adjusted behavior management techniques are used in order to prevent fainting, for example, applied tension (Vika et al. 2008)

ELIGIBILITY:
Inclusion Criteria:

* : school aged children (8 to10) years old. With or without previous dental experience

Exclusion Criteria:

* Medically compromised children. Refusal of participation.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children from 8 to 10 years with or without previous dental experience
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of intraoral injection fear | immediate
  self reported fear of intraoral injection through filling of a 12 questions of Intraoral Injection Fear scale, the scale has scores from 12 to 60 and the cut off score is 38, Below 38 is better as it means the child is not fearful from intraoral injections.

SECONDARY OUTCOMES:
Prevalence of dental fear | immediate
  children fear survey subscale

OTHER OUTCOMES:
Dental avoidance | immediate
  single question

CONTACTS AND LOCATIONS:
Overall Officials: Pediatric dentistry department, Study Chair — Faculty of oral and dental medicine

REFERENCES:
- [Background] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259
- [Background] Vika M, Raadal M, Skaret E, Kvale G. Dental and medical injections: prevalence of self-reported problems among 18-yr-old subjects in Norway. Eur J Oral Sci. 2006 Apr;114(2):122-7. doi: 10.1111/j.1600-0722.2006.00335.x. PMID 16630303
- [Background] El-Housseiny AA, Alsadat FA, Alamoudi NM, El Derwi DA, Farsi NM, Attar MH, Andijani BM. Reliability and validity of the Children's Fear Survey Schedule-Dental Subscale for Arabic-speaking children: a cross-sectional study. BMC Oral Health. 2016 Apr 14;16:49. doi: 10.1186/s12903-016-0205-0. PMID 27079656
- [Background] Armfield JM, Heaton LJ. Management of fear and anxiety in the dental clinic: a review. Aust Dent J. 2013 Dec;58(4):390-407; quiz 531. doi: 10.1111/adj.12118. PMID 24320894
- [Background] Oliveira MA, Vale MP, Bendo CB, Paiva SM, Serra-Negra JM. Dental Fear Survey: a cross-sectional study evaluating the psychometric properties of the Brazilian Portuguese version. ScientificWorldJournal. 2014;2014:725323. doi: 10.1155/2014/725323. Epub 2014 Aug 11. PMID 25184153
- [Background] McGoldrick P, Levitt J, de Jongh A, Mason A, Evans D. Referrals to a secondary care dental clinic for anxious adult patients: implications for treatment. Br Dent J. 2001 Dec 22;191(12):686-8. doi: 10.1038/sj.bdj.4801270. PMID 11792115
- [Background] Marshman, Z., Noble, F., Rodd, H., 2018. 'Your teeth you are in control.' Dental Nursing 14, 292-293. doi:10.12968/denn.2018.14.6.292
- [Background] Mednick, L.M., Claar, R.L., 2012. Treatment of severe blood-injection-injury phobia with the applied-tension method: Two adolescent case examples. Clinical Case Studies. doi:10.1177/1534650112437405
- [Result] Berge KG, Agdal ML, Vika M, Skeie MS. High fear of intra-oral injections: prevalence and relationship to dental fear and dental avoidance among 10- to 16-yr-old children. Eur J Oral Sci. 2016 Dec;124(6):572-579. doi: 10.1111/eos.12305. Epub 2016 Sep 30. PMID 27689943